CLINICAL TRIAL: NCT00736385
Title: Hyperinsulinemia and Insulin Resistance in Nonalcoholic Fatty Liver Disease. Metformin for the Treatment of Nonalcoholic Fatty Liver Disease: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Metformin for the Treatment of Nonalcoholic Fatty Liver Disease (NAFLD)
Acronym: NAFLD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00006196; K23DK062116 (NIH)
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2016-12

CONDITIONS: Fatty Liver
Keywords: nonalcoholic fatty liver disease
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): Metformin XR (extended-release) 2000 mg daily
  Interventions: Drug: Glucophage (Metformin)
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucophage (Metformin) — metformin XR 2000 mg daily for 12 months
  Other Names: metformin; Glucophage XR (extended-release); Glumetza; Fortamet; Riomet
  Arms: Metformin
Drug: Placebo — placebo 2000 mg daily for 12 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if Metformin is safe and useful in the treatment of NAFLD.

DETAILED DESCRIPTION:
NAFLD is a poorly understood disease which may cause an enlarged liver, abnormal liver test results, and scarring of the liver. It may occur more often in people with obesity, high levels of cholesterol (blood fats), diabetes (high blood sugar), or the insulin resistance syndrome (where a person's body does not respond to the hormone insulin which helps keep blood sugar levels normal). Currently, no effective drug treatment for NAFLD exists. There is increasing evidence that NAFLD may be a condition due to a problem with metabolism (the way your body uses energy). Previous studies have shown that high glucose (sugar) levels may play an important role in the development of fatty liver disease. Medications that decrease your natural glucose level may reduce the amount of fat in the liver and, therefore, might be useful in the treatment of NAFLD. Metformin, a drug approved by the U.S. Food and Drug Administration (FDA) for use in patients with diabetes, has been shown to improve fatty liver in animals and in a small number of human beings.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven NAFLD, determined within 12 months of study initiation

Exclusion Criteria:

* > 20 grams of alcohol/day
* impaired oral glucose tolerance test
* known diagnosis of diabetes mellitus
* hepatitis C infection
* cirrhosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manal F Abdelmalek, MD, MPH, Principal Investigator — Duke University Medical Center, Department of Medicine, Division of Gastroenterology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 subjects signed consent to participate. 2 subjects were screen failures. 9 subjects were randomized.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 4 | 5
Completed | 2 | 2
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Metformin: Metformin XR 2000 mg daily
  Glucophage (Metformin): metformin XR 2000 mg daily for 12 months
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Study Endpoints Will Include Measurements of Insulin Sensitivity, Hepatic Insulin Clearance, and Altered Parameters of Lipid Metabolism, Changes in the Histological Features That Define NAFLD, and Quantitative Measurements of Visceral and Peripheral Fat.
Time Frame: 24 months
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Tests the Postulate That Metformin Will Improve Insulin Sensitivity in NAFLD. Also Test the Postulate That Improving IR (Insulin Resistance) With an Insulin Sensitizing Agent Will Improve Biochemical and Histological Features of NAFLD.
Time Frame: 24 months
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Determine if Metformin Improves the Altered Parameters of Lipid Metabolism as Compared to Placebo.
Time Frame: 24 months
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Measure the Differential Effects of IR and Lipid Metabolism on Peripheral Mononuclear Cell (PBMC) Inflammatory Response and the Associated Hepatocyte Mitochondrial Ultrastructure and Measures of Oxidative Stress
Time Frame: 24 months
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=4) | Placebo (N=5)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bradycardia Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=4) | Placebo (N=5)
Neck pain, low back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
arthritis (shoulder and neck ) (Musculoskeletal and connective tissue disorders) | 0 | 1 — x-ray diagnosed shoulder and neck arthritis
Sinus headache, sinus infection, cold (Infections and infestations) | 1 | 2
Rash and itching or redness (Skin and subcutaneous tissue disorders) | 0 | 2
Stomach cramping, diarrhea and vomitting (Gastrointestinal disorders) | 2 | 0
bluriness of vision (Eye disorders) | 0 | 1
Low energy and low mood (Psychiatric disorders) | 0 | 1
atrial fibrillation (Cardiac disorders) | 0 | 1
Tooth pain (Infections and infestations) | 0 | 1
gross bloody urine-renal stone (Renal and urinary disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Cut wound (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early due to difficulties with enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes